CLINICAL TRIAL: NCT04170738
Title: Brain Indices of Stimulant Treatment in Drug-Naive Youth at Risk for Substance Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeffrey Newcorn (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Newcorn, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 17-1321; 1R21DA046029-01A1 (NIH)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Conduct Disorder; Substance Abuse
Keywords: ADHD; substance abuse risk; Adderall; fMRI; ADHD Treatment; Medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Substance-Related Disorders | interventions — Adderall; SLI381

STUDY DESIGN:
Intervention Model Description: 3-week intervention with Adderall as treatment for ADHD among youth with ADHD + Conduct problems. Pre and post fMRI performed as the outcome measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adderall (Experimental): dosage = start at 0.25-0.50mg/kg, adjusted as necessary pills by mouth
  Interventions: Drug: Adderall

INTERVENTIONS:
Drug: Adderall — 3 weeks of Adderall
  Other Names: Dextroamphetamine-Amphetamine

SUMMARY:
Childhood ADHD and comorbid oppositional defiant disorder (ODD) and conduct disorder (CD) are considered risk factors for subsequent substance abuse, and youth with both ADHD and ODD/CD are at greatest risk.

However, the effects of treatment of ADHD with stimulant medications such as methylphenidate (MPH) and mixed amphetamine salts (MAS) on risk for substance abuse are poorly understood. The study team propose to use fMRI to study the effects of extended release mixed amphetamine salts (MAS-XR) in drug-naïve youth 7-12 years at low risk (i.e., ADHD only) and high risk (i.e., ADHD + ODD/CD) for substance abuse on the brain reward system, to better understand the potential impact of these medications on an aspect of brain functioning which is thought to underlie vulnerability to substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* General: pre-pubertal (e.g. Tanner stage 1 or 2)
* age 7-12 inclusive
* signed consent/assent
* parent communicates sufficiently in English
* Has ADHD as determined by parent interview
* ADHD-Rating Scale-5 total score (interview with parent) of 1.5 SD > age/sex norms
* Youth with CD or severe ODD: CD or ODD + 2 symptoms of CD

Exclusion Criteria:

* major neurological/medical illness
* history of head injury
* fetal exposure to alcohol/drugs;
* diagnosis of major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, generalized anxiety, social phobia, Tourette's Disorder, PTSD, autism spectrum disorder) current suicidal ideation or past history of suicide attempt
* Wechsler Abbreviated Scale of Intelligence (WASI) score <75; 7)
* current treatment with stimulants (prior or current treatment with non-stimulants is permitted, but participants must be off medication for 2 weeks at baseline; youth who had a past, brief stimulant medication exposure of no more than about a month, and not within the past 6 months may be included .)
* current or past alcohol/drug use (interview; urine toxicology)
* psychological or medical condition which precludes being in the scanner (e.g., claustrophobia, morbid obesity)
* metal in the body that cannot be removed
* visual disturbances that may impair task performance
* precocious puberty (e.g. Tanner stage >2).

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Iliyan Ivanov, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk: Children with ADHD and ODD/CD
- Low Risk: Children with ADHD only
Period: Overall Study
Arm/Group | High Risk | Low Risk
Started | 26 | 7
Completed | 11 | 7
Not Completed | 15 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk | Low Risk | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.00 (1.483) | 10.14 (1.345) | 9.44 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Full Scale IQ (FSIQ) [Mean (Standard Deviation); unit: units on a scale] — Full range from 40-160, higher score indicating better intellectual functioning
  units on a scale | 102.45 (12.003) | 107.29 (11.041) | 104.9 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in fMRI Measure
Description: Bold activation change within the reward system. The contrasts in blood-oxygenation levels (BOLD) in regions of interest (ROIs).
Time Frame: baseline and 3 weeks post intervention
Population: Participants who provided imaging data
Measure: Mean (Standard Deviation); unit: BOLD signal
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 7 | 6
BOLD signal
  Reward Outcome Post-Pre Low>High, Left Amygdala | -0.957100 (1.365781) | 0.572517 (0.712410)
  Reward Outcome Post-Pre Low>High, ACC | -0.139000 (1.288470) | 1.876717 (1.615755)
  Reward Outcome Post-Pre Low>High, Ventral Striatum | 0.853514 (0.475767) | -0.321983 (1.075986504)
  Reward Outcome Post-Pre Low>High, Ventrolateral Pre-Frontal Cortex (VLPFC) | 0.712514 (0.944126) | 0.460432 (0.744686)

2. Secondary Outcome: ADHD Rating Score (ADHD RS)
Description: Subscale for Inattention scores range from 0-27, Subscale scores for Hyper (H/I) range from 0-27. The total ADHD score sums to a score of 0-54. Higher indicates more severe ADHD symptomology, and there are norm ranges, with clinical thresholds set at 1.5 SD above the mean for sex and age.
Time Frame: Pretreatment, baseline and Post-Treatment, average 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 11 | 7
score on a scale
  ADHRS-total baseline | 43.18 (7.264) | 39.86 (13.057)
  ADHRS-total post Tx | 20.36 (13.677) | 12.71 (5.314)
  ADHRS-hyper baseline | 20.55 (5.298) | 19.71 (6.651)
  ADHRS-hyper post Tx | 10.09 (7.355) | 8.86 (3.805)
  ADHRS-InAtt baseline | 22.64 (3.906) | 20.14 (7.988)
  ADHRS- InAtt post Tx | 10.27 (7.016) | 8.86 (3.805)

3. Secondary Outcome: Total Dose of MAS-XR
Description: Open label trial of MAS XR with flexible dosing and a suggested target of at least 0.5mg/kg
Time Frame: average 2 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 11 | 7
mg | 1487.09 (2108.303) | 745.00 (594.636)

4. Secondary Outcome: Change in Clinical Global Impression - Improvement (CGI-I)
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
  Change in CGi post treatment as compared to baseline.
Time Frame: baseline and post treatment, average 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 11 | 7
score on a scale | 2.0 (0.632) | 2.00 (0.577)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Adverse Events collected using parent report
Arm/Group | High Risk | Low Risk
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04170738/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT04170738/ICF_001.pdf